CLINICAL TRIAL: NCT00394420
Title: A Telephone Quitline Intervention for Smoking Cessation Through the Emergency Department
Brief Title: Emergency Department Telephone Quitline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1321-03
Record Dates: First submitted 2006-10-31; First posted 2006-11-01 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2010-01

CONDITIONS: Tobacco Dependence
MeSH Terms: conditions — Tobacco Use Disorder

INTERVENTIONS:
Behavioral: Telephone Quitline

SUMMARY:
The purpose of this preliminary study was to evaluate the intervention completion rate among cigarette smokers enrolled through the Emergency Department (ED) in a tobacco quitline (QL) and to assess the feasibility of a randomized controlled trial assessing the efficacy of this intervention.

DETAILED DESCRIPTION:
This pilot study was a prospective, randomized, controlled, un-blinded study using a convenience sample of cigarettes smokers recruited through the ED.

Utilizing a computerized block randomization schedule, subjects were randomized in blocks of four to receive a proactive QL intervention through an established QL or a United States Public Health Service (USPHS) self-help manual. Proactive telephone counseling describes counseling that is initiated by a counselor rather than the subject. Both groups received strong advice to quit from study personnel.

Names and telephone numbers of patients randomized to the QL group were faxed to the QL which then initiated contact with the patient. Multiple contact attempts were made over the following week by telephone. Patients in the QL were instructed to call the QL if they had not been reached in one week. QL counseling involved an initial 45-minute telephone session followed by up to four 10 to 15 minute follow-up sessions around their identified quit date. QL patients not successfully contacted within one week of enrollment were sent a letter inviting them to call as well as information on strategies to help them quit.

ELIGIBILITY:
Inclusion Criteria:

* We enrolled patients aged 18 or older who reported current daily cigarette smoking for at least one year and who indicated an interest in attempting to quit smoking.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2003-09; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome was completion of the QL intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Nicola E. Schiebel, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States